CLINICAL TRIAL: NCT01878773
Title: Prostate Delineation During Radiation Treatment Planning for Prostate Cancer: Comparison of High Quality Volume Computerized Tomography With Conventional Tomography and Magnetic Resonance Imaging
Brief Title: Prostate Delineation: High Quality Volume CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 12-5229-CE
Record Dates: First submitted 2012-10-24; First posted 2013-06-17 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI scan; External beam radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Quality Volume CT Scan; MRI Scan (Other): Patients will have the High Quality volume CT scan immediately after their CT scan followed by MRI Scan.
  Interventions: Other: High Quality Volume CT Scan; MRI Scan

INTERVENTIONS:
Other: High Quality Volume CT Scan; MRI Scan — Patients will have the High Quality volume CT scan immediately after their CT scan followed by MRI scan.
  --------------------------------------------------------------------------------

SUMMARY:
This study will look at how feasible it is to use a certain type of Computed Tomography (CT) to scan prostate cancer, called a high quality volume CT scan. It is hoped that this technique will help doctors provide a higher-quality image of the prostate cancer, making it easier to plan the area that will be treated. Using this type of CT scan will also lessen the amount of time patients spend in the scanner.

This study will not offer patients a different treatment for their prostate cancer. Patients will receive the most appropriate standard treatment whether or not they are in this study.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Subjects undergoing radical external beam radiotherapy for prostate cancer
3. Ability to provide written informed consent

Exclusion Criteria:

1. Age ≤ 18 years
2. Subjects not suitable for MRI scanning
3. 3 usable image sets not obtained during treatment planning scans.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Using different scanning methods for patients undergoing radical external beam radiotherapy for prostate cancer to determine inter-observer variability in prostate gland delineation on the images. | 6 months

SECONDARY OUTCOMES:
Determine the concordance between delineators in identifying the prostate apex on the 2 CT image sets. MRI will be considered the "gold-standard" for identifying the prostate apex. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, The Princess Margaret, Toronto, Ontario, Canada